CLINICAL TRIAL: NCT00039403
Title: A Phase I Study Of UCN-01 In Combination With Gemcitabine In Unresectable Or Metastatic Pancreatic Carcinoma
Brief Title: UCN-01 and Gemcitabine in Treating Patients With Unresectable or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02468; DM01-553; U01CA062461 (NIH); CDR0000069380 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 7-hydroxystaurosporine; Gemcitabine

ARMS (1):
- Treatment (UCN-01, gemcitabine hydrochloride) (Experimental): Patients receive gemcitabine IV over 1-2 hours on days 1 and 8 followed by UCN-01 IV over 3 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Sequential dose escalation of UCN-01 is followed by sequential dose escalation of gemcitabine. Cohorts of 3-6 patients receive escalating doses of UCN-01 and then gemcitabine until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 6 patients are treated at the recommended phase II dose.
  Interventions: Drug: 7-hydroxystaurosporine; Drug: gemcitabine hydrochloride; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 7-hydroxystaurosporine — Given IV
  Other Names: UCN-01
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of combining UCN-01 with gemcitabine in treating patients who have unresectable or metastatic pancreatic cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. UCN-01 may help gemcitabine kill more cancer cells by making tumor cells more sensitive to the drug

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and toxicity profile of UCN-01 when given in combination with gemcitabine to patients with unresectable or metastatic adenocarcinoma of the pancreas.

II. To characterize the pharmacokinetic profiles of gemcitabine and UCN-01 when given in combination and to correlate various measurements of UCN-01 with intracellular concentrations.

III. To determine recommended doses of UCN-01 and gemcitabine in combination to be used in a planned subsequent phase II trial.

SECONDARY OBJECTIVES:

I. To record the frequency, extent, and duration of any tumor responses. II. To correlate serum alpha-1 acid glycoprotein (AGP) levels with UCN-01 pharmacokinetics and toxicity.

OUTLINE: This is a dose-escalation study.

Patients receive gemcitabine IV over 1-2 hours on days 1 and 8 followed by UCN-01 IV over 3 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Sequential dose escalation of UCN-01 is followed by sequential dose escalation of gemcitabine.

Cohorts of 3-6 patients receive escalating doses of UCN-01 and then gemcitabine until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 6 patients are treated at the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable or metastatic adenocarcinoma of the pancreas
* Unidimensionally measurable disease

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Tumor lesions in a previously irradiated area are not considered measurable
* No known brain metastases

  * Patients with signs or symptoms of CNS metastasis at any time during screening must have a negative CT scan or MRI of the brain
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No prior coronary artery disease
* No symptomatic cardiac dysfunction
* No prior myocardial infarction
* No active angina (even if controlled by medication)
* No positive stress test
* No uncontrolled arrhythmia
* Left ventricular ejection fraction at least 45%
* Patients with symptoms suggestive of coronary artery disease or arrhythmia must have no evidence of cardiac pathology
* No symptomatic pulmonary dysfunction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to UCN-01 or other study agents
* No insulin-dependent diabetes mellitus
* No other concurrent uncontrolled illness
* No ongoing or active infections
* No concurrent psychiatric illness
* No other active malignancy
* No other solid tumor within the past 5 years except neoplasia in situ or nonmelanomatous skin cancer
* No social situations that would preclude study compliance
* No concurrent over-the-counter biologics
* No concurrent growth factors during the first study course
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 2 prior chemotherapy regimens (e.g., gemcitabine and/or experimental agents) alone or in combination with radiotherapy as neoadjuvant or adjuvant therapy for resectable, unresectable, or metastatic disease
* See Chemotherapy
* At least 6 weeks since prior radiotherapy and recovered
* Prior radiotherapy directed only at the primary tumor bed allowed
* No prior radiotherapy to the mediastinum, pelvis, lower spine, or more than 20% of bone marrow
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior investigational agents
* Concurrent enrollment in non-therapy trials (e.g., quality of life) allowed
* No concurrent herbal remedies
* No concurrent treatment for another active malignancy
* No concurrent warfarin for anticoagulation
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity | Up to 4 years
Pharmacokinetic profiles | Weeks 1-6 for UCN-01 and weeks 1 and 4 for intracellular gemcitabine
Recommended phase II doses | 3 weeks

SECONDARY OUTCOMES:
Frequency, extent, and duration of any tumor responses | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Linus Ho, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States